CLINICAL TRIAL: NCT05945095
Title: The Effect of Chewing Gum After Cesarean Section on Gastrointestinal System Functions, Pain and Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Dilek Kaloglu Binici, Principal Investigator (PhD Research Nurse), Artvin Coruh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Gum after cesarean section
Record Dates: First submitted 2023-04-05; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Mothers; Cesarean Section Complications
Keywords: General anesthesia,; Sleep Quality; Chewing Gum, Pain,; Cesarean section,
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain

STUDY DESIGN:
Intervention Model Description: The sample size in similar studies was examined and it was determined that at least 30 mothers should be included in the experimental and control groups.
  Assignment of pregnant women to the experimental and control groups will be made using a simple random numbers table.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Gum chewing group
  Interventions: Other: Gum chewing group
- Control group (No Intervention): Routine care

INTERVENTIONS:
Other: Gum chewing group — The mothers in the experimental group, on the other hand, will chew sugar-free gum for at least 15 minutes, starting from the second hour after the surgery.
  Arms: Experimental group

SUMMARY:
The study will be conducted on mothers who had planned cesarean section.After the birth, the information about the surgery in the personal information form will be completed. Then, mothers in the control group will be given standard postpartum care. The mothers in the experimental group, on the other hand, will chew sugar-free gum for at least 15 minutes, starting from the second hour after the surgery. The gum chewing process will be repeated every two hours. Mothers will be mobilized at the 8th sat after the birthday.

Pain levels of mothers in both groups will be evaluated every two hours after delivery.

In addition, the amount of analgesic use will be compared and comments will be made on the level of pain. The sleep quality of the postpartum women will be questioned the day after the cesarean section.

DETAILED DESCRIPTION:
The study will be conducted on mothers who had planned cesarean section. The sample size in similar studies was examined and it was determined that at least 30 mothers should be included in the experimental and control groups.

Assignment of pregnant women to the experimental and control groups will be made using a simple random numbers table.

In the data collection process of the research, the "personal information form" consisting of 24 questions and developed by the researchers as a result of the literature review, the "Richard-Campbell Sleep Scale" and the "Visual Comparison Scale (VAS)" will be used.

Prenatal interviews will be conducted with the pregnant women and their status of meeting the following inclusion criteria will be evaluated, and all pregnant women who comply with the criteria and agree to participate in the study will be asked questions regarding the prenatal period in the personal information form.

After the birth, the information about the surgery in the personal information form will be completed.

Then, mothers in the control group will be given standard postpartum care. The mothers in the experimental group, on the other hand, will chew sugar-free gum for at least 15 minutes, starting from the second hour after the surgery.

The gum chewing process will be repeated every two hours. Mothers will be mobilized at the 8th sat after the birthday. Pain levels of mothers in both groups will be evaluated every two hours after delivery.

In addition, the amount of analgesic use will be compared and comments will be made on the level of pain.

The sleep quality of the postpartum women will be questioned the day after the cesarean section.

Gastrointestinal system functions will be followed in the postoperative period and will be evaluated by asking questions about gas output and defecation time in the personal information form.

After the mothers in both groups have defecated, the data collection process will be completed from the mother concerned.

The data obtained will be entered into the SPSS (Statistical Package for the Social Sciences) 22.0 package program and evaluated with appropriate statistical analysis.

Inclusion Criteria for Research:

be 18 years or older, having a planned cesarean section, to receive general anesthesia during surgery, chronic constipation and no history of diarrhea be at least a primary school graduate, and is not a communication problem.

ELIGIBILITY:
Inclusion Criteria:

* Be eighteen years of age or older,
* Having a planned cesarean section,
* To receive general anesthesia in the surgery,
* No history of chronic constipation and diarrhea,
* At least primary school graduate
* Communication is not a problem.
* Exclusion Criteria:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 60 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-12-27 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | "change" is being assessed. up to 10-12 hours after cesarean section
  VAS is used to measure perceived pain. VAS is a 10cm line with anchor statements on lower end (no pain) and on upper end (extreme pain). The mother is asked to mark their current pain level on the line

SECONDARY OUTCOMES:
Richard-Campbell Sleep Scale (RCUI) | in the morning the day after the cesarean section
  The Turkish validity and reliability study of the scale, which was developed by Richards in 1987, was carried out by Özlü and Özer in 2015.
  Each item of the six-item scale, which evaluates the depth of night sleep, the duration of falling asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep and the noise level in the environment, is evaluated on a chart between 0-100 using the visual analog scale technique.
  A score of "0-25" from the scale indicates very bad sleep, and a score of "76-100" indicates very good sleep.
  The total score of the scale is evaluated over 5 items, and the sixth item, which evaluates the noise level in the environment, is excluded from the total score evaluation.
  As the score of the scale increases, the sleep quality of the patients also increases.
  The Cronbach's alpha value of the scale is 0.91.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek KALOĞLU BİNİCİ, PhD, Principal Investigator — Artvin Coruh University
Locations (1):
- Artvin State Hospital, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pereira Gomes Morais E, Riera R, Porfirio GJ, Macedo CR, Sarmento Vasconcelos V, de Souza Pedrosa A, Torloni MR. Chewing gum for enhancing early recovery of bowel function after caesarean section. Cochrane Database Syst Rev. 2016 Oct 17;10(10):CD011562. doi: 10.1002/14651858.CD011562.pub2. PMID 27747876